CLINICAL TRIAL: NCT04407260
Title: The Use of Oxygen Hoods in Patients Failing on Conventional High-flow Oxygen Delivery Systems, the Effects on Oxygenation, Mechanical Ventilation and Mortality Rates in Hypoxic Patients With COVID-19. A Prospective Controlled Cohort Study.
Brief Title: Use of Oxygen Hoods in Patients Failing on Conventional High-flow Oxygen Delivery Systems, Effects on Oxygenation in Hypoxic COVID-19 Patients. Prospective Cohort Study.
Status: Completed | Type: Observational
Sponsor: Northwell Health (Other)
Responsible Party: Principal Investigator, David Dayya, Attending Physician, Northwell Health
Other Study IDs: HoodStudy701
Record Dates: First submitted 2020-05-27; First posted 2020-05-29 (Actual); Last update posted 2022-12-02 (Actual); Status verified 2022-11

CONDITIONS: COVID -19; Respiratory Failure; Hypoxia
MeSH Terms: conditions — COVID-19; Respiratory Insufficiency; Hypoxia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (2):
- Intervention: Patients on oxygen hoods who have fail conventional high-flow oxygen delivery systems.
  Interventions: Device: Oxygen Hood
- Control: Patients maintained on conventional high-flow oxygen delivery systems (such as non-rebreather masks, high-flow nasal cannula, BiPAP, CPAP) or who have failed on these conventional symptoms and were subsequently mechanically ventilated.

INTERVENTIONS:
Device: Oxygen Hood — High-Flow Oxygen Hood with neck dam and intake and exhaust tubing incorporating a Bacterial/Viral HEPA filter and optional PEEP attachment.
  Other Names: Oxygen Helmets
  Groups: Intervention

SUMMARY:
To determine whether the use of oxygen hoods as compared to conventional high-flow oxygen delivery systems, and the effects on oxygenation, mechanical ventilation and mortality rates in hypoxic patients with COVID-19.

DETAILED DESCRIPTION:
To determine whether Oxygen hoods improve O2-saturation (SaO2), and how they effect length of hospitalization, and in-hospital mechanical ventilation and mortality rates in Covid-19 patients when compared to conventional high-flow oxygen delivery systems. Oxy-hemoglobin saturation is continuously measured by pulse-oximetry including immediately before and after oxygen hood placement, and will be measured in controls.

Comparison/Control Group The control cohort includes COVID-19 patients presenting for treatment prior to 4/3/20 when hyperbaric oxygen hoods were not available. Patients maintained on, or those failing on conventional O2- delivery systems and subsequently receiving mechanical ventilation will be studied.

All patients included must have tested positive using PCR swabs and/or been diagnosed based on clinical/laboratory standard diagnostic criteria. Medical management will include evolving treatment regimens and other standard medical treatments widely used at time of study in all hypoxic COVID-19 patients.

Prognostic/confounding covariates are to be collected through Electronic Medical Record (EMR) chart review and compared between intervention and control cohorts. including: Age, Body Mass Index (BMI), Gender, Chronic Lung disease - COPD, Asthma (CLD), cardiovascular disease - CAD, CHF, Chronic Dysrhythmia (CVD), chronic kidney disease (CKD), Immunosuppression - History of Cancer, Immunosuppressive medication, HIV (Immunosuppression), Diabetes Mellitus (DM), and pertinent lab markers.

Routine follow-up evaluation is maintained until final in-hospital outcomes are known including:

1. Oxygen Difference pre/post-hood (SaO2 difference, %)
2. Intubation/MV status (Intubated)
3. Survival/Mortality (Expired)
4. Hospital Length of Stay (LOS, days)

Randomization/Blinding Randomization is not possible as it is unethical to deny a hypoxic patient an alternative approved means of oxygenation for patients failing on conventional oxygen delivery systems. No blinding of participants or investigators.

ELIGIBILITY:
Inclusion Criteria

* Hospital census is reviewed for ALL patients seen in the Emergency Department admitted with COVID -19 diagnosis and experiencing hypoxia requiring supplemental high-flow oxygen delivery or who have required mechanical ventilation.
* Consent (native language services provided).
* No limitations/restrictions on age, sex, race/ethnicity, comorbidities, pregnancy status, DNR/DNI status.

Exclusion Criteria

* SaO2 > 90% on conventional high-flow O2-delivery system.
* Confinement anxiety post-oxygen hood placement with request for removal.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All COVID-19 patients presenting to the hospital prior to the availability of oxygen hoods were reviewed for eligibility and assignment to the control cohort.
  All COVID-19 patients presenting to the hospital after the availability of oxygen hoods were reviewed for eligibility and assignment to the intervention cohort if they were failing on conventional high-flow oxygen delivery systems.
Sampling Method: Non-Probability Sample
Enrollment: 136 (Actual)
Dates: Start 2020-03-06 (Actual); Primary Completion 2020-05-01 (Actual); Study Completion 2020-05-01 (Actual)

PRIMARY OUTCOMES:
Oxygen saturation | 3/6/2020 - 5/1/2020
  Continuous pulse oximetry monitoring
In-hospital Intubation/Mechanical Ventilation Status | 3/6/2020 - 5/1/2020
  Intubation/mechanical Ventilation at any point during hospitalization.
In-hospital Mortality | 3/6/2020 - 5/1/2020
  In-hospital Mortality status
Length of Hospitalization | 3/6/2020 - 5/1/2020
  Duration of hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: David Dayya, DO, PhD, MPH, Principal Investigator — Phelps Hospital - Northwell Health; Owen J O'Neill, MD, MPH, Principal Investigator — Phelps Hospital - Northwell Health
Locations (1):
- Phelps Hospital, Sleepy Hollow, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided
If other researchers are investigating similar research question will consider sharing IPD.

REFERENCES:
- [Background] Organization WH. Rolling updates on Coronavirus disease (COVID - 19) - Coronavirus disease (COVID-19) Situation Report.: World Health Organization, 2020.
- [Background] Control CfD. Recommended Preparedness and Response Activities in Healthcare. Supplement C: Preparedness and Response In Healthcare Facilities. Public Health Guidance for Community-Level Preparedness and Response to Severe Acute Respiratory Syndrome (SARS) Version 2/3.
- [Background] Richardson S, Hirsch JS, Narasimhan M, Crawford JM, McGinn T, Davidson KW; the Northwell COVID-19 Research Consortium; Barnaby DP, Becker LB, Chelico JD, Cohen SL, Cookingham J, Coppa K, Diefenbach MA, Dominello AJ, Duer-Hefele J, Falzon L, Gitlin J, Hajizadeh N, Harvin TG, Hirschwerk DA, Kim EJ, Kozel ZM, Marrast LM, Mogavero JN, Osorio GA, Qiu M, Zanos TP. Presenting Characteristics, Comorbidities, and Outcomes Among 5700 Patients Hospitalized With COVID-19 in the New York City Area. JAMA. 2020 May 26;323(20):2052-2059. doi: 10.1001/jama.2020.6775. PMID 32320003
- [Background] Berlin DA, Gulick RM, Martinez FJ. Severe Covid-19. N Engl J Med. 2020 Dec 17;383(25):2451-2460. doi: 10.1056/NEJMcp2009575. Epub 2020 May 15. No abstract available. PMID 32412710
- [Background] Health. NDo. Amid Ongoing COVID-19 Pandemic, Governor Cuomo Announces State Department of Health Has Approved New Protocol to Allow BiPAP Machines to be Converted Into Ventilators.
- [Background] Wang L, He W, Yu X, Hu D, Bao M, Liu H, Zhou J, Jiang H. Coronavirus disease 2019 in elderly patients: Characteristics and prognostic factors based on 4-week follow-up. J Infect. 2020 Jun;80(6):639-645. doi: 10.1016/j.jinf.2020.03.019. Epub 2020 Mar 30. PMID 32240670
- [Background] Patel BK, Wolfe KS, Pohlman AS, Hall JB, Kress JP. Effect of Noninvasive Ventilation Delivered by Helmet vs Face Mask on the Rate of Endotracheal Intubation in Patients With Acute Respiratory Distress Syndrome: A Randomized Clinical Trial. JAMA. 2016 Jun 14;315(22):2435-41. doi: 10.1001/jama.2016.6338. PMID 27179847
- [Background] Patel BK, Wolfe KS, MacKenzie EL, Salem D, Esbrook CL, Pawlik AJ, Stulberg M, Kemple C, Teele M, Zeleny E, Macleod J, Pohlman AS, Hall JB, Kress JP. One-Year Outcomes in Patients With Acute Respiratory Distress Syndrome Enrolled in a Randomized Clinical Trial of Helmet Versus Facemask Noninvasive Ventilation. Crit Care Med. 2018 Jul;46(7):1078-1084. doi: 10.1097/CCM.0000000000003124. PMID 29595563
- [Background] K M. Oxygen Administration: What Is the Best Choice? Respiratory Therapy 2015.
- [Background] Department of Health and Human Services - Food and drug Administration - Conference of CDRH OoDEO. Device Evaluation and Approval., 2002.
- [Background] UN-TBftLDC. Local production could solve shortages of essential pandemic-fighting equipment., 2020.
- [Background] MEDICINE. ECFH. ECHM position on Hyperbaric Oxygen Therapy (HBOT) in multiplace hyperbaric chambers during coronavirus disease (COVID-19) outbreak.
- [Background] B L, A C, Z B, et al. COVID-19: Oxygen Escalation Therapy and Noninvasive Ventilation. EmDocs 2020. http://www.emdocs.net/covid-19-oxygen-escalation-therapy-and-noninvasive-ventilation/ (accessed April 15, 2020).
- [Background] Prevention CfDCa. Evaluating and Testing Persons for Coronavirus Disease 2019 (COVID-19). 2020.
- [Background] Ashraf-Kashani N, R K. High-flow nasal oxygen therapy. BJA Education;17(2):57-62.
- [Background] Rengasamy S, Shaffer R, Williams B, Smit S. A comparison of facemask and respirator filtration test methods. J Occup Environ Hyg. 2017 Feb;14(2):92-103. doi: 10.1080/15459624.2016.1225157. PMID 27540979
- [Background] Marini JJ, Gattinoni L. Management of COVID-19 Respiratory Distress. JAMA. 2020 Jun 9;323(22):2329-2330. doi: 10.1001/jama.2020.6825. No abstract available. PMID 32329799
- [Background] IBM SPSS Statistics for Windows [program]. 25.0 version. Armonk, NY: IBM Corp., Released 2017.
- [Derived] Dayya D, O'Neill OJ, Feiertag TD, Tuazon-Boer R, Sullivan J, Perez L, Gurash S, Eaton M, Bodley T, Marker J, Smykowski E, Hall T. The use of oxygen hoods in patients failing on conventional high-flow oxygen delivery systems, the effects on oxygenation, mechanical ventilation and mortality rates in hypoxic patients with COVID-19. A Prospective Controlled Cohort Study. Respir Med. 2021 Apr;179:106312. doi: 10.1016/j.rmed.2021.106312. Epub 2021 Feb 12. PMID 33636568